CLINICAL TRIAL: NCT06641934
Title: Current Survey on Chemotherapy-Related Myelosuppression and Clinical Management in Chinese County-level Tumor Patients
Status: Not yet recruiting | Type: Observational
Sponsor: The First Affiliated Hospital of Xinxiang Medical College (Other)
Collaborators: Xinxiang Central Hospital of Henan province (Unknown); Linzhou People Hospital (Unknown); Inner Huang County Traditional Chinese Hospital (Unknown); Changyuan People Hospital (Unknown); Huojia County People Hospital (Unknown); Huojia County Alliance Hospital (Unknown); Qinyang People Hospital (Unknown); Xinan County People Hospital (Unknown); Henan Hongli Hospital (Unknown); Army Hospital of the 83rd Army (Unknown); Anyang Cancer Hospital (Unknown); Puyang Hospital of Traditional Chinese Medicine (Unknown); Puyang Huimin Hospital (Unknown); Hebi People Hospital (Unknown); The Second People Hospital of Xinxiang Henan (Unknown)
Responsible Party: Sponsor
Other Study IDs: CHASE009; Renco Quick Review No. (19) (Other: FirstAffiliatedHXinxiangMC)
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Myelosuppression
Keywords: Myelosuppression
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Chemotherapy-Related Myelosuppression: Chemotherapy-Related Myelosuppression Clinical Management
  Interventions: Other: No intervention; Observational study
- Chemotherapy-related myelosuppression, primary prevention, treatment rate and clinical management: Chemotherapy-related myelosuppression, primary prevention, treatment rate and clinical management
  Interventions: Other: No intervention; Observational study
- Chemotherapy-induced myelosuppression, secondary prevention, treatment rates, and clinical managemen: no intervention
  Interventions: Other: No intervention; Observational study

INTERVENTIONS:
Other: No intervention; Observational study — No intervention

SUMMARY:
Current Survey on Chemotherapy-Related Myelosuppression and Clinical Management in Chinese County-level Tumor Patients

DETAILED DESCRIPTION:
The purpose of this research project was to gain an in-depth understanding of the myelosuppression of cancer patients in counties in China after receiving chemotherapy-based treatment regimens through a cross-sectional survey with the help of an online questionnaire system, and to investigate doctors' cognition and treatment concepts of chemotherapy-induced myelosuppression. 1. Fill the gaps in relevant domestic research and provide basic data for follow-up longitudinal studies and intervention studies; 2. Analyze the influencing factors and coping strategies of chemotherapy-induced bone marrow suppression from multiple perspectives, so as to provide reference for improving the knowledge level and treatment level of patients and doctors; 3. Provide more scientific guidance and suggestions for chemotherapy for cancer patients, help patients reduce the harm of bone marrow suppression, improve the survival rate and quality of life of patients, and also provide strong data support for the prevention and treatment of tumors and promote the development of cancer prevention and treatment.

ELIGIBILITY:
Inclusion Criteria：

* The confirmed malignant tumor is one of the non-small cell lung cancer/small cell lung cancer/breast cancer/gastric cancer/esophageal cancer/colorectal cancer/gynecological malignant tumor (ovarian cancer, cervical cancer, endometrial cancer).
* Patients who need to receive chemotherapy in the past 3 months and should continue to receive chemotherapy in the future
* The relevant diagnosis and treatment information involved in the survey is complete: only patients with at least 1-2 examination results after 1 week after chemotherapy can be included
* Understand and sign the informed consent form
* The chemotherapy regimen received for the most recent chemotherapy should be one of the following

  1. Non-small cell lung cancer TP scheme NP scheme DP scheme EP scheme GP scheme AP scheme Docetaxel/pemetrexed monotherapy Gemcitabine monotherapy Tigio monotherapy ADCs Other monotherapy or combination regimens containing platinum or taxane drugs Drug regimens that combine the above chemotherapy regimens (e.g., immunosuppressants, targeted therapy drugs, etc.)
  2. Small cell lung cancer with etoposide-containing combination regimens Platinum-containing combination regimens (except etoposide) Monotherapy or combination regimen containing topotecan, gemcitabine, paclitaxel Drug regimens that combine the above chemotherapy (e.g., immunosuppressants, targeted therapy drugs, etc.)
  3. reast cancer ddEC sequential T regimen Anthracyclines and taxanes: TAC, TE, EC-T, ddEC-T, FEC-T regimens Combined taxane protocols: TP, AP, TC, Anthracycline combination regimen: EC, FEC Taxane monotherapy Yew combined with platinum Other platinum-containing regimens: NP, GP ADC drugs Microtubule inhibitors: NVB, taxanes (nab-paclitaxel, paclitaxel liposome, docetaxel), eutidrone, eribulin Microtubule inhibitors in combination with capecitabine Anthracycline monotherapy Drug regimens that combine the above chemotherapy (e.g., targeted therapy drugs, etc.)
  4. Gastric cancer SOX protocol XELOX scheme FOLFOX protocol DCF scheme ADCs Other monotherapy or combination regimens containing platinum or taxanes or fluorouracil Drug regimens that combine the above chemotherapy (e.g., immunosuppressants, targeted therapy drugs, etc.)
  5. Esophageal cancer taxane + platinum regimen CF protocol DCF scheme FOLFOX protocol XELOX scheme FLOT scheme FOLFIRI PROTOCOL ECF protocol ECX scheme EOF scheme EOX protocol Other monotherapy or combination regimens containing platinum or taxane or fluorouracil Drug regimens that combine the above chemotherapy (e.g., immunosuppressants, targeted therapy drugs, etc.)
  6. COLORECTAL CANCER FOLFOXIRI FOLFOX FOLFIRI XELOX Other monotherapy or combination regimens containing platinum or fluorouracil or raltitrexed Drug regimens that combine the above chemotherapy (e.g., immunosuppressants, targeted therapy drugs, etc.)
  7. Gynecologic malignancies:platinum + taxane or its combination regimen Monotherapy or combination chemotherapy containing docetaxel/gemcitabine/topotecan/irinotecan Regimens (except platinum + taxanes) Other monotherapy or combination chemotherapy regimens containing platinum, taxanes, or anthracyclines

Exclusion Criteria：

* Patients with concurrent chemoradiotherapy,
* Patients with sequential chemoradiotherapy, and the irradiation site of radiotherapy is flat bone, sternum, and pelvis;
* Patients with active bleeding before or during treatment; If the patient has received targeted drugs such as CDK4/6 inhibitors or chidaaniline in the front-line treatment, which have a great impact on the blood phase, the drug can be discontinued for at least half a month before it can be included
* Patients who, in the opinion of other physicians, would cause non-chemotherapy-related myelosuppression

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Chinese County-level Tumor Patients
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-10-20 (Estimated); Primary Completion 2025-10-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Incidence of chemotherapy-related myelosuppression and current status of prophylactic therapy | 2024.09-2025.09
  The incidence and treatment status of chemotherapy-related myelosuppression were investigated in the form of questionnaires Like what：
  1. Did bone marrow suppression occur after the previous cycle of chemotherapy? (First chemotherapy/occurrence/non-occurrence)
  2. Did CIM (chemotherapy-induced myelosuppression) occur during this chemotherapy? (Multiple selections allowed)
  3. Survey questions about existing CIM therapeutic drugs

SECONDARY OUTCOMES:
Incidence of chemotherapy-related myelosuppression | 2024.09-2025.09
  Through questionnaire survey：the incidence of neutropenia during chemotherapy treatment and the rate of primary and secondary prophylaxis;
the rate and economic burden of neutropenia treatment during chemotherapy treatment | 2024.09-2025.09
  Through questionnaire survey：the rate and economic burden of neutropenia treatment during chemotherapy treatment like what:Is there an additional financial burden? A.<500 yuan, B.500-<1000 yuan, C.1000-<3000 yuan, D.≥3000 yuan
the incidence of thrombocytopenia and the rate of primary and secondary prevention and treatment during chemotherapy treatment | 2024.09-2025.09
  Through questionnaire survey： the incidence of thrombocytopenia and the rate of primary and secondary prevention and treatment during chemotherapy treatment like what:Is there primary /secondary prevention in this chemotherapy? Yes/No
thrombocytopenia treatment rate and economic burden during chemotherapy treatment | 2024.09-2025.09
  Through questionnaire survey： thrombocytopenia treatment rate and economic burden during chemotherapy treatment like what：Does it increase the financial burden of patients to a certain extent? Yes/No
the incidence and treatment rate of anemia during chemotherapy treatment; | 2024.09-2025.09
  Through questionnaire survey：the incidence and treatment rate of anemia during chemotherapy treatment like what:Extensive-stage small cell lung cancer/advanced non-small cell lung cancer/advanced HR-negative breast cancer/advanced gastric cancer/advanced esophageal cancer/advanced colorectal cancer/advanced gynaecological malignancy, the overall incidence of CIM in patients with chemotherapy is approximately ()? What is the incidence of grade ≥ 3 ()? A.<10% B. 10%-24% C. 25%-49% D,≥50%
Long and/or short acting granulocyte colony-stimulating factor (G-CSF) and/or Chinese patent medicine usage rate and application scenario cost analysis | 2024.09-2025.09
  Through questionnaire survey：Long and/or short acting granulocyte colony-stimulating factor (G-CSF) and/or Chinese patent medicine usage rate and application scenario cost analysis like what:The number of patients on G-CSF prophylaxis ________ digits/month A. ≤20 B. 21-49 C. 50-99 D. ≥100 What is the proportion of patients with total chemotherapy (including chemotherapy combined with other treatments)________% A. 0%-25% B. 26%-49% C. 50%-75% D. 75%-100% Number of patients with neutropenia afterG-CSF prophylaxis _______ position/month A. ≤20 B. 21-49 C. 50-99 D. ≥100 What percentage of patients are treated with G-CSF prophylaxis________% A. 0%-25% B. 26%-49% C. 50%-75% D. 75%-100%
Recombinant human interleukin-11 and/or thrombopoietin (TPO) and/or thrombopoietin receptor agonists (TPO-RA) and/or cost analysis of application scenarios | 2024.09-2025.09
  Through questionnaire survey：Recombinant human interleukin-11 and/or thrombopoietin (TPO) and/or thrombopoietin receptor agonists (TPO-RA) and/or cost analysis of application scenarios like what:Number of patients receiving chemotherapy (including chemotherapy in combination with other treatments), the number of patients given terbiao/roprostim/other prophylaxis: _______ places/month, A. ≤ 20 B. 21-49 C. 50-99 D. ≥100 What is the proportion of patients with total chemotherapy (including chemotherapy combined with other treatments)________% A. 0%-25% B. 26%-49% C. 50%-75% D. 75%-100% Number of patients with thrombocytopenia after administration of terbiao/roprostim pre/other prophylaxis _______ place/month A. ≤20 B. 21-49 C. 50-99 D. ≥100 What percentage of patients given TPIAO/roprostim prophylaxis ________% A. 0%-25% B. 26%-49% C. 50%-75% D. 75%-100%
Erythropoietin and/or iron and/or Chinese patent medicine usage rate and application scenario cost analysis | 2024.09-2025.09
  Through questionnaire survey：Erythropoietin and/or iron and/or Chinese patent medicine usage rate and application scenario cost analysis like what:What kind of drug treatment to use (multiple choices are allowed)A.Red blood cell transfusion B.Erythropoietin C.Hematopoietic raw materials such as iron supplementation D.Traditional Chinese medicine treatment E.No treatment requiredF. Other: Please describe: ________________

CONTACTS AND LOCATIONS:
Overall Officials: Ji YH yinghua, Dr., Study Chair — The First Affiliated Hospital of Xinxiang Medical College
Locations (1):
- The First Affiliated Hospital of Xinxiang Medical College, Xinxiang, Henan, China

IPD SHARING:
Plan to Share IPD: Undecided